CLINICAL TRIAL: NCT03141528
Title: Self-learning Versus Instructor-led Learning in Basic Life Support Training - A Randomized Controlled Trial
Brief Title: Self-learning vs Instructor-led Learning in BLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Req-2016-00071
Record Dates: First submitted 2017-02-09; First posted 2017-05-05 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Basic Life Support
Keywords: Self-learning; Instructor-led learning; Long-term retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instructor-led learning (Active Comparator): This group will train their technical CPR-skills with supervision by a tutor (either general practitioner or medical student, all trained in CPR teaching)
  Interventions: Other: Instructor-led learning
- Self-learning (Experimental): This group will Train alone without supervision and without communicating with the other participants.
  Interventions: Other: Self-learning

INTERVENTIONS:
Other: Self-learning — Training without supervision
  Arms: Self-learning
Other: Instructor-led learning — Supervision by a tutor (either general practitioner or medical student, all trained in CPR teaching)
  Arms: Instructor-led learning

SUMMARY:
This study investigates whether there is a difference in the BLS skills in first year medical students directly after training and three months later, when randomly assigned to self-learning versus instructor-led training courses.

DETAILED DESCRIPTION:
This is a randomized controlled trial investigating whether self-learning versus instructor-led learning results in the same BLS skills in first year medical students directly after training and three months later.

When participants attend the "Erweiterte Erste Hilfe für Studierende der Humanmedizin" they will receive a short introduction about the study. The investigators will invite all first year students to participate in the study. As the study is voluntarily, participants need to sign a written informed consent. After that, the investigators will randomize the students to either group A or Group B. Group A will train their technical CPR-skills with supervision by a tutor (either general practitioner or medical student, all trained in CPR teaching) and group B will train without supervision. The participants in group B will not be allowed to communicate with each other during the training and they will be prevented from watching each other. The training will take about 30 minutes for each group. Directly after the training each group will be tested and the printed report form from the Laerdal Skill Reporter will be obtained for each participant. In the test the students will perform CPR in a simulated scenario as a first responder. The scenario is: "A male person has collapsed at the railway station." The participant should start CPR as learned in the training. During the CPR a departmental research fellow will observe the study participants and record BLS/AED actions on a scoring sheet.

The investigators will record three cycles of two minutes CPR (with five times 30:2 compression : ventilation intervals, as recommended by the current international resuscitation guidelines). During the three cycles an AED will be delivered and the study participant has to apply the AED and deliver a shock - after three cycles the study terminates.

After the BLS/AED competence testing, both groups will continue the rest of their first aid course together and the first part of the study ends. Three months later, the investigators will repeat the same scenario over the same time interval and record the same parameters. At the end of the second testing, a short feedback will be provided on the BLS/AED competence and further practice will be provided to the students to improve their CPR competence. From this point forward no further data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* First year medical students at the University of Bern participating in the course "Erweiterte Erste Hilfe für Studierende der Humanmedizin" with written informed consent.

Exclusion Criteria:

* Students with professional BLS-experience, unable to perform BLS, or missing informed consent will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD, Principal Investigator — University Hospital Bern Inselspital
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Instructor-led Learning | Self-learning
Started | 122 | 118
Completed | 75 | 77
Not Completed | 47 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Instructor-led Learning | Self-learning | Total
Number analyzed (Participants) | 122 | 118 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 118 | 240
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21 [20 to 22] | 21 [20 to 22] | 21 [20 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 69 | 141
  Male | 50 | 49 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 122 | 118 | 240
Region of Enrollment [Number; unit: participants]
  Switzerland | 122 | 118 | 240

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correct Compressions
Description: The percentage of correct compressions obtained from the printed report from the Laerdal Skill Reporter.
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: percentage of correct compressions
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
percentage of correct compressions
  Teaching | 48 [10 to 83] | 42 [14 to 81]
  Follow - up | 28 [6 to 59] | 47 [12 to 78]

2. Secondary Outcome: Assessment of the Participants BLS Competences After Test
Description: Assessment of the participant's BLS competence by the study team after test.
  Rated on a Visual Analogue Scale from 0-100mm, where 0mm = completely incompetent, no idea what to do, and 100mm = totally competent, cannot be done better.
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 122 | 118
units on a scale
  Teaching | 73 [61 to 81] | 68 [56 to 77]
  Follow-up | 68 [56 to 81] | 65 [54 to 77]

3. Secondary Outcome: Self-assessment of the Participants BLS Competences Before Test
Description: The participants assessment of their own BLS competences. Rated on a Visual Analogue Scale from 0-100mm, where 0mm = completely incompetent, no idea what to do, and 100mm = totally competent, cannot be done better.
Time Frame: before first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 122 | 118
score on a scale
  Teaching | 71 [63 to 77] | 70 [63 to 80]
  Follow-up | 60 [49 to 70] | 59 [49 to 68]

4. Secondary Outcome: Assessment of the Teaching Method
Description: The participants assessment of the teaching method. Rated on a Visual Analogue Scale from 0-100mm, where 0mm = completely inefficient, and 100mm = totally efficient, nothing can be done better."
Time Frame: after first BLS course
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 122 | 118
score on a scale | 80 [70 to 90] | 75 [62 to 84]

5. Secondary Outcome: Average Ventilation Volume
Description: Ventilation volume from the printed report from the Laerdal Skill Reporter (LSR)
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
ml
  Teaching | 790 [640 to 1010] | 810 [620 to 1150]
  Follow-up | 615 [530 to 770] | 660 [570 to 800]

6. Secondary Outcome: Number of Ventilations Per Minute
Description: Number of ventilations per minute from the printed report from the Laerdal Skill Reporter (LSR)
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: (ventilations/min)
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
(ventilations/min)
  Teaching | 2 [2 to 3] | 2 [2 to 3]
  Follow-up | 2 [2 to 3] | 3 [2 to 3]

7. Secondary Outcome: Percentage of Correct Ventilations
Description: Percentage of correct ventilations from the printed report from the Laerdal Skill Reporter (LSR)
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: percentage of corrent ventilations
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
percentage of corrent ventilations
  Teaching | 25 [5 to 50] | 22 [3 to 50]
  Follow-up | 50 [15 to 71] | 41 [17 to 70]

8. Secondary Outcome: Number of Participants Using Correct Ratio of Compressions:Ventilations
Description: the relationship between ventilations and compressions from the printed report from the Laerdal Skill Reporter (LSR). Ventilations - relationship 30 compressions and 2 ventilations.
Time Frame: after first BLS course and 3 months later
Measure: Count of Participants; unit: Participants
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
Participants
  Teaching | 18 | 16
  Follow-up | 6 | 8

9. Secondary Outcome: Compression Depth
Description: Compression depth from the printed report from the Laerdal Skill Reporter (LSR)
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
mm
  Teaching | 52 [44 to 57] | 52 [45 to 57]
  Follow-up | 50 [42 to 56] | 53 [46 to 58]

10. Secondary Outcome: Number of Compressions Per Minute
Description: Number of compressions per minute from the Laerdal Skill Reporter (LSR)
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: compressions per minute
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
compressions per minute
  Teaching | 54 [46 to 58] | 51 [44 to 57]
  Follow-up | 57 [53 to 64] | 59 [51 to 63]

11. Secondary Outcome: Compression Frequency
Description: Compression frequency from the Laerdal Skill Reporter (LSR). Compressions per minute ventilation break included.
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: compressions per minute
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
compressions per minute
  Teaching | 112 [105 to 118] | 111 [103 to 116]
  Follow - up | 113 [104 to 121] | 114 [103 to 122]

12. Secondary Outcome: Compressions Too Shallow
Description: Total percentage of Compressions too shallow from the Laerdal Skill Reporter (LSR)
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: percentage of Compressions too shallow
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
percentage of Compressions too shallow
  Teaching | 25 [4 to 82] | 24 [2 to 76]
  Follow-up | 44 [3 to 87] | 18 [4 to 66]

13. Secondary Outcome: False Hand Placement During Compressions
Description: False hand placement during compressions.
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: percentage of False hand placement durin
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
percentage of False hand placement durin
  Teaching | 6 [0.3 to 20] | 6 [0 to 34]
  Follow-up | 13 [0. to 41] | 15 [0 to 96]

14. Secondary Outcome: Incomplete Decompression
Description: Incomplete decompression from the Laerdal Skill Reporter (LSR)
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: percentage of Incomplete decompression
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 105 | 105
percentage of Incomplete decompression
  Teaching | 0 [0 to 0.3] | 0 [0 to 0.3]
  Follow - up | 0 [0 to 0] | 0 [0 to 0]

15. Secondary Outcome: Time From Start of Test Till Call for Help
Description: Time measured from the beginning of the test until the participant calls for help.
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 122 | 118
seconds
  Teaching | 10 [7 to 16] | 12 [8 to 18]
  Follow-up | 9 [5 to 16] | 8 [5 to 15]

16. Secondary Outcome: Time From Start of Test Till First Compression
Description: Time measured from the beginning of the test until the participant makes the first compression.
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 122 | 118
seconds
  Teaching | 35 [27 to 46] | 35 [26 to 46]
  Follow-up | 28 [23 to 35] | 25 [21 to 32]

17. Secondary Outcome: Time From Start of Test Till First Ventilation
Description: Time measured from the beginning of the test until the participant makes the first ventilation.
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 122 | 118
seconds
  Teaching | 70 [56 to 112] | 64 [55 to 92]
  Follow-up | 93 [56 to 106] | 63 [45 to 97]

18. Secondary Outcome: Time From Start of Test Till First Shock
Description: Time measured from the beginning of the test until the participant gives the first shock.
Time Frame: after first BLS course and 3 months later
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Instructor-led Learning | Self-learning
Number analyzed (Participants) | 122 | 118
seconds
  Teaching | 100 [82 to 120] | 118 [95 to 145]
  Follow-up | 83 [73 to 102] | 88 [75 to 107]

ADVERSE EVENTS:
Time Frame: 2 Hours
Description: No Adverse Event possible. The Study were only performed on Manikins.
Arm/Group | Instructor-led Learning | Self-learning
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/188
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/118
Other Adverse Events (participants affected / at risk) | 0/122 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT03141528/Prot_SAP_000.pdf